CLINICAL TRIAL: NCT06061159
Title: The ED95 of Single Intravenous Bolus Remimazolam Besylate in Pediatric Patients During General Anesthesia Induction:a Randomised,Double-blind Clinical Trial
Brief Title: The ED95 of Single Intravenous Bolus Remimazolam Besylate in Pediatric Patients During General Anesthesia Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAHoWMU-CR2023-03-107
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Pediatric; ED95; Sedation; General Anesthesia
Keywords: remimazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1-3years old (Experimental): single intravenous bolus remimazolam about 5min before general anesthesia induction
  Interventions: Drug: Remimazolam besylate
- 3-6years old (Experimental): single intravenous bolus remimazolam about 5min before general anesthesia induction
  Interventions: Drug: Remimazolam besylate
- 6-12years old (Experimental): single intravenous bolus remimazolam about 5min before general anesthesia induction
  Interventions: Drug: Remimazolam besylate

INTERVENTIONS:
Drug: Remimazolam besylate — initial dose is 0.2mg/kg；adjust dosage is 0.05mg/kg
  Other Names: single intravenous bolus remimazolam according to biased coin design
  Arms: 6-12years old
Drug: Remimazolam besylate — initial dose is based on the findings from the school-age group；adjust dosage is 0.05mg/kg
  Other Names: single intravenous bolus remimazolam according to biased coin design
  Arms: 1-3years old; 3-6years old

SUMMARY:
Due to the incomplete development of systems and low pain thresholds in the pediatric population, good general anesthesia is required during the perioperative period to ensure the smooth progress of the surgery.Propofol is often used for anesthesia induction in clinical work, which can achieve good anesthesia effects. However, this drug has obvious injection pain and is prone to significant inhibition of blood circulation, and may even lead to adverse conditions such as respiratory depression in children. For the pediatric population, maintaining appropriate anesthesia depth and stable circulation during the induction period of general anesthesia has always been a focus of attention and research by anesthesiologists.Remimazolam besylate is a new type of water-soluble ultra short acting benzodiazepine drug that is hydrolyzed and metabolized by plasma esterase in the body, independent of liver and kidney function, and the metabolite zolam propionic acid has no pharmacological activity; Rapid onset and failure, short sedation recovery time; Has little impact on respiration and circulation; And there is no injection pain.Remazolam besylate is highly suitable for children due to its characteristics, and some studies have demonstrated the safety of intravenous injection of Remazolam besylate. However, there is limited research on its dosage exploration, which to some extent limits its clinical application in children.This study aims to explore the 95% effective dose (ED95) of single intravenous injection of remidazolam besylate in children of different age groups, providing a theoretical basis for the use of remidazolam besylate in pediatric anesthesia.

DETAILED DESCRIPTION:
This experiment was divided into three groups based on the age of the children, namely 1-3 years old, 4-6 years old, 7-12 years old, with an initial dose of 0.2mg/kg. The time of consciousness loss in the children was evaluated after injection of ramazolam besylate to determine whether sedation had been achieved. The next dose was adjusted to 0.05mg/kg according to biased coin design,to further explore the ED95 of a single intravenous injection of ramazolam in children of different age groups.

ELIGIBILITY:
Inclusion Criteria:

1. with American Society of Anesthesiologists (ASA) physical status I or II；
2. aged 1-12 years；
3. children with weight for age within the normal range；
4. were scheduled general anesthesia surgery

Exclusion Criteria:

1. Children who had gastrointestinal,Cardiovascular or endocrine dysfunction;
2. contraindication to preoperative sedation or had a known allergy or hypersensitive reaction to remimazolam;
3. recently respiratory infection, mental disorder;
4. other reasons that researchers hold it is not appropriate to participate in this trial.

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2024-02-27 (Actual); Study Completion 2024-02-27 (Actual)

PRIMARY OUTCOMES:
the time of the loss of consciousness(LOC) | during anaesthetic induction
  Modified Observers Assessment of Alertness/Sedation (MOAA/S) score of 1 or deeper within 1 minute, and maintained until the end of the 5-minute observation period.

SECONDARY OUTCOMES:
Modified observer's assessment of alertness／sedation（MOAA/S）scale | Every 1 minutes after single intravenous bolus remimazolam
  5-Subject responds readily to name spoken in a normal tone; 4 -Lethargic response of a subject to a name spoken in a normal tone; 3 -The subject responds only after a name is called loudly and repeatedly; 2 -The subject responds only after mild prodding or shaking;
  1 -The subject responds only after a painful trapezius squeeze; 0 -The subject does not respond to painful trapezius squeeze. MOAA/S score ≤ 1 points represent successful sedation
BIS | Every 1 minutes after single intravenous bolus remimazolam
  BIS values range from 0 to 100. A value of 0 represents the absence of brain activity, and 100 represents the awake state.
  BIS values between 60 to 80 represent sedation; BIS values between 40 to 60 represent adequate general anesthesia for a surgery; values less than 40 represent a deep hypnotic state.
Recovery time | Within up to 30 minutes after child's first eye opening in the postoperative period
  The time from discontinuation of sevoflurane to the first open eye of the children and to achieve the modified aldrete scole ≥9.
  then the aldrete scole's minimum value is 0 and maximum value is 10, and higher scores mean a better or outcome.
  The modified aldrete scole consists of five items. Each item is scored 0-2 yielding a total between 0 and 10.
Number of children with adverse effects | Up to 24 hours including preoperative, intraoperative, and postoperative periods
  Number of children with adverse effects:
  １、Bradycardia and/or hypotension need for hemodynamic support; 2、Desaturation is defined as Oxygen desaturation <90%; 3、Nausea and vomiting; 4、Any adverse effects requiring interventions.
Rate of Pediatric anesthesia emergence delirium | Within up to 15-30 minutes after child's first eye opening in the postoperative period
  The pediatric anesthesia emergence delirium scale consists of five items. Each item is scored 0-4 yielding a total between 0 and 20.
  The degree of emergence delirium increased directly with the total score. pediatric anesthesia emergence delirium scale ≥12 at any time indicates presence of emergence delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Huacheng Liu, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Yuhang Cai, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University; Leqi Dong, Principal Investigator — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- The second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

REFERENCES:
- [Derived] Cai YH, Dong LQ, Zhong JW, Lin Z, Chen CD, Zhu LB, Lin XK, Szmuk P, Liu HC. ED50 and ED95 of remimazolam for loss of consciousness in young children: a dose-finding study for induction of anaesthesia. Br J Anaesth. 2025 Jun;134(6):1709-1716. doi: 10.1016/j.bja.2025.02.004. Epub 2025 Mar 18. PMID 40107902